CLINICAL TRIAL: NCT00823303
Title: A Phase 4 Randomized Multicenter Open Label Trial of Paricalcitol Versus Calcitriol for Efficacy and Safety in Stage 3 or 4 Ckd Patients With Secondary Hyperparathyroidism
Brief Title: Paricalcitol Versus Calcitriol for Efficacy and Safety in Stage 3/4 Chronic Kidney Disease (CKD) With Secondary Hyperparathyroidism (SHPT)
Acronym: PACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Henry Ford Hospital (Other); Northwestern University Feinberg School of Medicine (Other); Endeavor Health (Other); Abbott (Industry)
Responsible Party: Principal Investigator, Daniel W. Coyne, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22095
Record Dates: First submitted 2008-12-12; First posted 2009-01-15 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease
Keywords: PTH; Active Vitamin D; hypercalcemia; Chronic Kidney Disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Hypercalcemia | interventions — paricalcitol; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paricalcitol (Experimental): titrated to achieve 40-60% PTH suppression
  Interventions: Drug: Paricalcitol
- Calcitriol (Active Comparator): titrated to achieve 40-60% PTH suppression
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Paricalcitol — 1 mcg daily, adjusted to achieve 40-60% PTH suppression
  Other Names: Zemplar
  Arms: Paricalcitol
Drug: Calcitriol — 0.25 mcg daily, adjusted to achieve 40-60% PTH suppression
  Other Names: Rocaltrol
  Arms: Calcitriol

SUMMARY:
Secondary Hyperparathyroidism (SHPT) occurs in many patients with kidney disease and leads to bone disease. Active forms of vitamin D, calcitriol and paricalcitol, treat SHPT, but may have different effects on blood calcium. This study will randomize patients with SHPT and stage 3 or 4 CKD to treatment with calcitriol or paricalcitol, and monitor patients for the incidence of high blood calcium, and effectiveness of SHPT treatment.

DETAILED DESCRIPTION:
General Design

* Open label, active comparator, multicenter, parallel group, phase 4 study of paricalcitol versus calcitriol for suppression of PTH in stage 3 and 4 CKD patients with SHPT.
* Total study duration is 26 weeks (1 week screening, 24 weeks active medications, 1 week follow up.
* Patients meeting inclusion/exclusion criteria including baseline laboratory results will be randomized to paricalcitol or calcitriol, and enter a 24 weeks treatment phase. Visits, including safety and efficacy laboratory tests will be at weeks 4, 8, 12, 18, and 24. A follow up visit will be performed 1 week after stopping study medication.

ELIGIBILITY:
Inclusion Criteria

1. Age >18; Able to give informed consent
2. Chronic kidney disease, and estimated GFR 15 to 60 ml/min using the abbreviated MDRD equation
3. intact PTH (iPTH) >120 pg/ml at baseline
4. albumin corrected calcium > 8.5 mg/dL to < 10.0 mg/dL at baseline
5. Phosphorus < 4.6 mg/dL at baseline
6. If on a phosphorus binder; no change in dose within the 4 weeks prior to screening

Exclusion Criteria

1. Receiving any active form of vitamin D within 4 weeks prior to screening (calcitriol, doxercalciferol; paricalcitol; alfacalcidol)
2. Receiving >50,000 IU per month of ergocalciferol or > 1000 IU of cholecalciferol per day within the previous 30 days.
3. history of primary HPT
4. On prednisone > 30 days within the previous 6 months
5. receiving bisphosphonates or calcitonin within the previous 12 months
6. Non-elective hospitalization within the previous 30 days.
7. Expected to initiate dialysis or receive a kidney transplant within the next 6 mo.
8. History of renal or other organ transplant
9. History of parathyroidectomy or previous diagnosis of primary hyperparathyroidism
10. Receiving cinacalcet within 4 weeks prior to screening.
11. An active drug/alcohol dependence or abuse history
12. History of non-compliance with visits or medications that preclude study compliance in the opinion of the investigator
13. Pregnant, or able to become pregnant and unwilling to use a birth control method considered reliable by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-02; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Coyne, MD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University, St Louis, Missouri

REFERENCES:
- [Result] Coyne DW, Goldberg S, Faber M, Ghossein C, Sprague SM. A randomized multicenter trial of paricalcitol versus calcitriol for secondary hyperparathyroidism in stages 3-4 CKD. Clin J Am Soc Nephrol. 2014 Sep 5;9(9):1620-6. doi: 10.2215/CJN.10661013. Epub 2014 Jun 26. PMID 24970869

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paricalcitol | Calcitriol
Started | 54 | 56
Completed | 45 | 45
Not Completed | 9 | 11

BASELINE CHARACTERISTICS:
Population: Stage 3 and 4 CKD with SHPT, age >18, a stable dose of phosphate binder (if receiving a binder), estimated glomerular filtration rate (eGFR) of 15-59 mL/min using the abbreviated MDRD equation, PTH >120 pg/mL, albumin-corrected calcium >8.5 mg/dL and <10.0 mg/dL, phosphorus <4.6 mg/dL.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol | Calcitriol | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (13.2) | 64.7 (12.6) | 65.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 30 | 54
  Male | 30 | 26 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 41 | 74
  White | 18 | 14 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Hypercalcemia
Description: Serum Calcium 10.5 mg/dL or higher, confirmed by repeat measurement.
Time Frame: 24 week treatment period
Measure: Number; unit: participants
Arm/Group | Paricalcitol | Calcitriol
Number analyzed (Participants) | 53 | 54
participants | 3 | 1
Statistical Analysis 1: Comparison: Paricalcitol vs Calcitriol; Test type: Non-Inferiority or Equivalence — On the basis of prior published reports, we estimated a 5% rate of hypercalcemia with paricalcitol and a 30% rate with calcitriol. To have a 90% power to detect a difference at the P=0.05 confidence level, 42 patients per group were needed. Assuming a 30% dropout rate over the course of the study, we planned to randomize 110 patients; p = 0.36, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Paricalcitol | Calcitriol
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/54
Other Adverse Events (participants affected / at risk) | 15/53 | 12/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paricalcitol (N=53) | Calcitriol (N=54)
Hypercalcemia (Endocrine disorders) | 0 (0) | 1 (1) — Hypercalcemia requiring or prolonging hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paricalcitol (N=53) | Calcitriol (N=54)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 15 (15) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No